CLINICAL TRIAL: NCT01770288
Title: Psychophysical Aspects of Maximal Anaerobic Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: University of Haifa (Other); Zinman College of Physical Education and Sports Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 8-12
Record Dates: First submitted 2013-01-06; First posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Anaerobic Performance
Keywords: Anerobic exercise; Pain; Analgesia; Diffuse Noxious Inhibitory Control (DNIC); psychological stress
MeSH Terms: conditions — Pain; Agnosia; Stress, Psychological

ARMS (1):
- Anaerobic Performance (Experimental)
  Interventions: Other: Anaerobic wingate test

INTERVENTIONS:
Other: Anaerobic wingate test

SUMMARY:
During anaerobic exercise, the metabolic pathway of glycolysis is used in order to produces high-energy compounds adenosine triphosphate (ATP).The level of lactic acid in the blood is a marker to the increased protons concentration and acidosis.nevertheless, the increased level of protons in addition to the release of bradykinin causes pain during the exercise that limited the subject's performance. Therefore, it is assumed that the individual pain sensitivity might determine the subject's performance.

Aims: To investigate the role of the DNIC efficiency in prediction of anaerobic performance in humans (2) to study the role of peripheral pro-nociceptive processing in mediating pain during anaerobic exercise and its contribution to the subjects' performance (3) to assess the function of pain-related psychological factors in anaerobic performance.

DETAILED DESCRIPTION:
To the best of our knowledge, no study has investigated the balance between the endogenous anti-nociceptive properties of the individual and the anaerobic-evoke pro-nociceptive activity in determining the maximal performance during anaerobic exercise. Moreover, the interaction between psychological factors and pro- and anti- nociceptive processes that are operated during anaerobic exercise, need to be investigated.

Methods: Forty healthy men and women, between the ages of 18-40 will be involved in the study. Each participant will complete 3 psychological questionnaires regarding their personality traits: Pain Catastrophizing Scale (PCS), State-Trait Anxiety Inventory and Perceived Stress Questionnaire. Pain psychophysics tests will be used for evaluating the individual pain perception, prior and subsequent to the anaerobic exercise: (1) DNIC will be tested using a paradigm of two remote noxious stimuli with one, the 'conditioning stimulus' (immersing the hand in tub containing 8°c water), inhibiting the other, the 'test pain' (pressure pain threshold) in order to assess the endogenous analgesia (EA) efficiency (2) heat and pressure pain thresholds, and (3) temporal summation of painful heat and mechanical stimuli that reflect the neuroplasticity of the central nervous system following peripheral noxious stimulation. In addition, Anaerobic performance will be evaluated during Wingate test,and blood lactate will be measured. Gene related pain ill be tested using saliva samples .

ELIGIBILITY:
Inclusion Criteria:

healthy Volunteers

Exclusion Criteria:

pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Pain psychophysics tests | 1 year
  DNIC will be tested using a paradigm of two remote noxious stimuli with one, the 'conditioning stimulus' (immersing the hand in tub containing 8°c water), inhibiting the other, the 'test pain' (pressure pain threshold) in order to assess the EA efficiency (2) heat and pressure pain thresholds, and (3) temporal summation of painful heat and mechanical stimuli that reflect the neuroplasticity of the central nervous system following peripheral noxious stimulation.

SECONDARY OUTCOMES:
Lactate concentration | 1 year
  Lactate concentration at rest will be measures using a portable lactate analyzer
The anaerobic performance | 1 year
  will be evaluated during executing of Wingate test

CONTACTS AND LOCATIONS:
Overall Officials: Einat Kodesh, PhD, Principal Investigator — University of Haifa
Locations (1):
- Zinman College for Physical Education and Sport Sciences at the Wingate Institute, Netanya, Israel